CLINICAL TRIAL: NCT05181852
Title: A Randomised, Double Blind, Placebo Controlled Study to Investigate the Pharmacodynamic Effects of IP2015 in Healthy Male Subjects Using the Intradermal Capsaicin Model
Brief Title: Study to Investigate the Pharmacodynamic Effects of IP2015 in Healthy Male Subjects Using the Intradermal Capsaicin Model
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Initiator Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IP2015CS03
Record Dates: First submitted 2021-11-20; First posted 2022-01-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Drug Evaluation; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IP2015_dose 1 (Experimental): Active
  Interventions: Drug: IP2015, dose 1
- IP2015_dose 2 (Experimental): Active
  Interventions: Drug: IP2015, dose 2
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Pregabalin (Active Comparator): Comparator
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: IP2015, dose 1 — Active
  Other Names: Test drug
  Arms: IP2015_dose 1
Drug: IP2015, dose 2 — Active
  Other Names: Test drug
  Arms: IP2015_dose 2
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Pregabalin — Comparator
  Other Names: Comparator
  Arms: Pregabalin

SUMMARY:
This is a Phase I, randomised, double-blind, placebo-controlled, 4-way crossover study to investigate the PD effects, safety, tolerability and PK/PD correlation of two single oral dose levels of IP2015 compared to 300 mg pregabalin and placebo in healthy male subjects using the ID capsaicin model.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male, with a skin type compatible with capsaicin measurements.
* Healthy as determined by a responsible physician, based on medical evaluation including medical history, physical examination, concomitant medication, vital signs, 12-lead ECG, clinical laboratory evaluations.
* Subject must be in good general health with a skin type compatible with the measures, and without significant skin allergies, pigmentary disorders, or any active dermatological conditions that might interfere with the conduct of the study.

Exclusion Criteria:

* Any significant CNS, cardiac, pulmonary, metabolic, renal, hepatic (including Gilbert's syndrome), gastrointestinal (GI) or psychiatric conditions, or history of fainting or syncope or such condition that, in the opinion of the Investigator, may place the subject at an unacceptable risk as a participant in the study, may interfere with the interpretation of safety or tolerability data obtained in this study, or may interfere with the absorption, distribution, metabolism or excretion (ADME) of drugs, or with the completion of treatment according to this Protocol.
* Clinically relevant history of abnormal physical or mental health interfering with the study as determined by medical history and physical examinations obtained during Screening as judged by the Investigator (including [but not limited to], neurological, psychiatric, endocrine, cardiovascular, respiratory, GI, hepatic, or renal disorder).
* Clinically relevant abnormal laboratory results (including hepatic and renal panels, complete blood count, chemistry panel and urinalysis), 12-lead ECG and vital signs, or physical findings at Screening. In case of uncertain or questionable results, tests performed during Screening may be repeated to confirm eligibility or judged to be clinically irrelevant for healthy subjects.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-01-05 (Estimated); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain related assessments of effect | A 6 hours time interval after dosing
  The area of hyperalgesia

SECONDARY OUTCOMES:
Pain related assessments of effect | A 6 hours time interval after dosing
  Subjective rating of pain
Pain related assessments of effect | A 6 hours time interval after dosing
  Pain VAS score of hyperalgesia
Pain related assessments of effect | A 6 hours time interval after dosing
  Area and pain VAS score of brush-evoked allodynia
Pain related assessments of effect | A 6 hours time interval after dosing
  Area of flare (AF)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Connell, MD, Principal Investigator — MAC UK

IPD SHARING:
Plan to Share IPD: No